CLINICAL TRIAL: NCT00760396
Title: A Placebo-Controlled, Ascending Multiple-Dose Study to Evaluate the Safety and Pharmacokinetics of VGX-1027 in Healthy Subjects
Brief Title: Multiple-Dose Study of VGX-1027 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VGX Pharmaceuticals, LLC (Industry)
Collaborators: GeneOne Life Science, Inc. (Industry)
Responsible Party: C. Jo White, MD, VGX Pharmaceuticals, Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CAT002
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Healthy
Keywords: healthy volunteers
MeSH Terms: interventions — 3-phenyl-4,5-dihydro-5-isoxazole acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): 40mg QD dose group
  Interventions: Drug: VGX-1027
- Group 2 (Experimental): 100mg QD dose group
  Interventions: Drug: VGX-1027
- Group 3 (Experimental): 200mg QD dose group
  Interventions: Drug: VGX-1027
- Group 4 (Experimental): 200mg BID dose group
  Interventions: Drug: VGX-1027

INTERVENTIONS:
Drug: VGX-1027 — Subjects will

SUMMARY:
The purpose of this study is to evaluate the safety profile, tolerability and pharmacokinetics following multiple oral doses of 40mg to 200mg VGX 1027 in healthy subjects administered for 5 days.

DETAILED DESCRIPTION:
This study will evaluate:

* The safety and tolerability of multiple oral doses of VGX 1027 in the range of 40 to 400mg.
* The pharmacokinetics of VGX 1027 in healthy subjects following the first oral dose (Day 1) and at steady state (Day 5).

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent.
* Healty subjects as determined by no clinically significant deviation from normal as judged by the investigator in medical history, physical examination, ECGs and clinical laboratory evaluations.
* Body Mass Index (BMI) of 18 to 30kg/m2 ±0.5kg/m2 inclusive.

Exclusion Criteria:

* Women who are of childbearing potential.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or prior to study drug administration.
* Male subjects who are unwilling to agree to practice barrier contraception during study participation and 3 months following dosing.
* Any significant acute or chronic medical illness
* Current or recent (within 3 months) gastrointestinal disease that may impact the absorption of the drug.
* Any major surgery within 4 weeks of enrollment.
* Donation of blood or plasma to a blood bank or in a clinical study (except a screening visit) within 4 weeks of enrollment.
* Blood transfusion within 4 weeks of enrollment.
* Inability to tolerate oral medication.
* Inability to be venipunctured and/or tolerate venous access.
* Recent (within 6 months) drug or alcohol abuse.
* History of bleeding disorder.
* History of head trauma or seizures.
* Any other sound medical, psychiatric and/or social reason as determined by the Investigator.
* Evidence of organ dysfunction or any clinically significant deviation from normal in vital signs, physical examination, ECG, or clinical laboratory determination.
* Positive urine screen for drugs of abuse
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen, HIV 1/2 antibody
* History of any significant drug allergy
* Exposure to any investigational druge within 4 weeks prior to enrollment or greater than 4 weeks for investigational drugs that may have a longer half life.
* Use of any prescription drugs, over the counter acid controllers within 4 weeks prior to enrollment.
* Use of any other drugs, including over the counter vitamins, medications and/or herbal preparations within 2 weeks prior to enrollment
* Use of oral, injectable or implantable hormonal contraceptive agents within three months prior to enrollment
* Use of alcohol containing beverages within 1 week prior to enrollment
* Use of grapefruit containing products within 1 week prior to enrollment
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety as determined by vital signs, ECGs, clinical laboratory evaluations and AE reporting. | Day 8

SECONDARY OUTCOMES:
Pharmacokinetics | Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Stephan A Bart, MD, Principal Investigator — SNBL Clinical Pharmacology Center, Inc.
Locations (1):
- SNBL Clinical Pharmacology Center, Inc., Baltimore, Maryland, United States